CLINICAL TRIAL: NCT00054392
Title: A Randomized, Phase III Multicenter Trial Of Gemcitabine In Combination With Carboplatin Or Paclitaxel Plus Carboplatin In Patients With Metastatic (Stage IIIB, IV) Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Stage IIIB, Stage IV, or Recurrent Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Not opened at Fox Chase Cancer Center
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: ALPHA-A1-99002L; CDR0000270434 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Lung Cancer
Keywords: adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; large cell lung cancer; recurrent non-small cell lung cancer; squamous cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Carboplatin; Gemcitabine; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as gemcitabine, carboplatin, and paclitaxel use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which chemotherapy regimen is more effective in treating non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of different combination chemotherapy regimens in treating patients who have stage IIIB, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with stage IIIB or IV or recurrent non-small cell lung cancer treated with gemcitabine and carboplatin vs gemcitabine and paclitaxel vs paclitaxel and carboplatin.
* Compare the overall response rate and time to progression in patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to weight loss within the past 6 months (less than 5% vs at least 5%), disease stage (IIIB vs IV), and brain metastases (present vs absent). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and carboplatin IV over 15-30 minutes on day 1.
* Arm II: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and paclitaxel IV over 3 hours on day 1.
* Arm III: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 15-30 minutes on day 1.

In all arms, treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every 6 weeks during study treatment, and then every 3 months until progressive disease is documented.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 1,134 patients (378 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC) of 1 of the following types:

  * Squamous cell
  * Adenocarcinoma
  * Large cell anaplastic
  * Bronchoalveolar
  * Non-small cell carcinoma not otherwise specified NOTE: Mixed tumors are categorized by the predominant cell type (tumors with small-cell anaplastic elements are ineligible)
* Evidence of at least 1 of the following:

  * Clinically documented recurrent disease after prior radiation or surgery
  * Stage IV disease (distant metastases)
  * Stage IIIB disease presenting with 1 of the following:

    * Pleural or pericardial effusion by CT scan or chest x-ray
    * Pleural implants documented pathologically or seen on CT scan or x-ray
* Measurable or evaluable disease
* No brain metastases unless clinically stable after surgery and/or radiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* AST less than 5 times upper limit of normal

Renal

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 40 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No hypersensitivity to agents that contain Cremophor EL (polyoxyethylated castor oil)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for advanced NSCLC

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy
* No prior radiotherapy to the only site of measurable disease, unless the site had subsequent progression of disease documented by physical exam, radiography, or pathology
* No concurrent radiotherapy (except for brain metastases)

Surgery

* See Disease Characteristics

Other

* No concurrent aminoglycoside antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-09; Primary Completion 2001-09 (Actual); Study Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
Tumor response rate
Time to disease progression
Quality of life as measured by the Functional Assessment of Cancer -Lung (FACT-L) questionnaire at baseline, every 6 weeks during study treatment, and then every 3 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Treat, MD, Study Chair — Fox Chase Cancer Center
Locations (57):
- United States (57):
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - New Hope Cancer and Research Institute - Pomona, Pomona, California
  - Lawrence and Memorial Hospital, New London, Connecticut
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - Cancer Center of Indiana, New Albany, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Annapolis Oncology Center, Annapolis, Maryland
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Fallon Clinic at Worcester Medical Center, Worcester, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Howell Township, New Jersey
  - Jersey Shore Cancer Center at Jersey Shore University Medical Center, Neptune City, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Mercer Bucks Oncology-Hematology, Trenton, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Cape Fear Valley Medical Center, Fayetteville, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Falling Spring Medical Associates, Chambersburg, Pennsylvania
  - Hematology-Oncology Associates of Northeastern Pennsylvania, Dunmore, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Richard G. Laube Cancer Center at ACMH, Kittanning, Pennsylvania
  - Lancaster Cancer Center, Lancaster, Pennsylvania
  - Central Pennsylvania Hematology and Medical Oncology Associates, PC, Lemoyne, Pennsylvania
  - Paoli Hematology-Oncology PC at Paoli Memorial Hospital, Paoli, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Drexel University College of Medicine - Center City Hahnemann Campus, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center CCOP Research Base, Philadelphia, Pennsylvania
  - Pennsylvania Oncology Hematology Associates, Incorporated - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Coastal Cancer Center - Myrtle Beach, Myrtle Beach, South Carolina
  - Family Cancer Center, PLLC - Collierville, Collierville, Tennessee
  - Baptist Regional Cancer Center at Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - University of Virginia Cancer Center at UV Health System, Charlottesville, Virginia
  - David Lee Outpatient Cancer Center at Charleston Area Medical Center, Charleston, West Virginia
  - Morgantown Internal Medicine Group, Incorporated, Morgantown, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia

REFERENCES:
- [Result] Edelman MJ, Belani CP, Socinski MA, Ansari RH, Obasaju CK, Chen R, Monberg MJ, Treat J; Alpha Oncology Research Network. Outcomes associated with brain metastases in a three-arm phase III trial of gemcitabine-containing regimens versus paclitaxel plus carboplatin for advanced non-small cell lung cancer. J Thorac Oncol. 2010 Jan;5(1):110-6. doi: 10.1097/JTO.0b013e3181c59a3a. PMID 20035187
- [Result] Obasaju CK, Ansari RH, Socinski MA, Chen R, Monberg MJ, Catalano RB, Marinucci DM, Liles DK, Ribeiro MJ, Comis RL, Treat J; Alpha Oncology Research Network. A Comparison of white and African American outcomes from a three-arm, randomized, phase III multicenter trial of advanced or metastatic non-small cell lung cancer. J Thorac Oncol. 2010 Jul;5(7):993-1000. doi: 10.1097/jto.0b013e3181e29cf3. PMID 20593535
- [Result] Treat JA, Gonin R, Socinski MA, Edelman MJ, Catalano RB, Marinucci DM, Ansari R, Gillenwater HH, Rowland KM, Comis RL, Obasaju CK, Belani CP; Alpha Oncology Research Network. A randomized, phase III multicenter trial of gemcitabine in combination with carboplatin or paclitaxel versus paclitaxel plus carboplatin in patients with advanced or metastatic non-small-cell lung cancer. Ann Oncol. 2010 Mar;21(3):540-547. doi: 10.1093/annonc/mdp352. Epub 2009 Oct 15. PMID 19833819
- [Result] Treat J, Edelman MJ, Belani CP, Socinski MA, Monberg MJ, Chen R, Obasaju CK; Alpha Oncology Research Network. A retrospective analysis of outcomes across histological subgroups in a three-arm phase III trial of gemcitabine in combination with carboplatin or paclitaxel versus paclitaxel plus carboplatin for advanced non-small cell lung cancer. Lung Cancer. 2010 Dec;70(3):340-6. doi: 10.1016/j.lungcan.2010.02.011. Epub 2010 Mar 27. PMID 20347506
- [Result] Treat J, Belani CP, Edelman MJ, et al.: A randomized phase III trial of gemcitabine (G) in combination with carboplatin (C) or paclitaxel (P) versus paclitaxel plus carboplatin in advanced (Stage IIIB, IV) non-small cell lung cancer (NSCLC): update of the Alpha Oncology trial (A1-99002L). [Abstract] J Clin Oncol 23 (Suppl 16): A-LBA7025, 627s, 2005.